CLINICAL TRIAL: NCT02521519
Title: Short Term Effects of Medial Branch Block vs Para-spinal Injection in Muscle Patients With Non-specific Chronic Low Back Pain
Brief Title: Short Terms Effects of Medial Branch Block vs Para-spinal Muscle Injection in Patients With Non-specific CLBP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Yoram Shir, Director of the Alan Edwards Pain Management Unit, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 14-190
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain, Mechanical
Keywords: Facet induced pain; Myofascial pain; Trigger points; Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- One side of the patient's back (Other): medial branch block (MBB): Using sterile conditions, 25 gauge needles will be placed in the desired position. In its final position for the L3 and L4 vertebrae the needle tip should reside at the junction of the superior articular process and the transverse process. At the L5-S1 level the needle tip should reach the junction between the sacral ala and the superior articular process of S1. Following a negative aspiration 0.5ml of injectate will be injected into each site.
  Interventions: Other: Medial branch block in one side
- Other side of the patient's back (Other): These injections will target the deep para-spinal muscles between the spinous process and inter-pedicular line of the L3-5 vertebrae. Under fluoroscopic guidance, a 25-gauge needle will be advanced, directed towards the lamina at the mid-distance between inter-pedicular line and the spinous process of the L3, L4 and L5 vertebrae, until touching the bone. A straight forceps will be attached to the junction of the skin and the needle; the needle will then be withdrawn by 1.4cm, to reside inside the muscle bulk. A five ml syringe diameter will be used to point 1.4 cm withdrawal. Following a negative blood aspiration, each level will be injected with 0.5 ml of the injectate.
  Interventions: Other: paravertebral deep intramuscular (PDI) injection

INTERVENTIONS:
Other: Medial branch block in one side — MBB: Using sterile conditions, 25G needles will be placed in the desired position. In its final position for the L3 and L4 vertebrae the needle tip should reside at the junction of the superior articular process and the transverse process. At the L5-S1 level the needle tip should reach the junction between the sacral ala and the superior articular process of S1. Following a negative aspiration 0.5ml of injectate will be injected into each site.
  Arms: One side of the patient's back
Other: paravertebral deep intramuscular (PDI) injection — injections will target the deep para-spinal muscles between the spinous process and inter-pedicular line of the L3-5 vertebrae. Under fluoroscopic guidance, a 25-gauge needle will be advanced, directed towards the lamina at the mid-distance between inter-pedicular line and the spinous process of the L3, L4 and L5 vertebrae, until touching the bone. A straight forceps will be attached to the junction of the skin and the needle; the needle will then be withdrawn by 1.4cm, to reside inside the muscle bulk. A five ml syringe diameter will be used to point 1.4 cm withdrawal. Following a negative blood aspiration, each level will be injected with 0.5 ml of the injectate.
  Arms: Other side of the patient's back

SUMMARY:
This study compares the efficacy of medial branch block (MBB) vs. paravertebral deep intramuscular (PDI) injection for pain relief in chronic low back pain. Based on randomization in first intervention session, one side receives MBB and the other side takes PDI and in second session the pattern reverses.

DETAILED DESCRIPTION:
Pain relief following medial branch block (MBB) might be due to facet joints desensitization and/or myofascial trigger points' desensitization. Patients will be randomized to two groups. The first group receives MBB in one side and paravertebral deep intramuscular (PDI) injection in the other side of the back. Next week the pattern of injection will be reversed so the side which had received MBB will take PDI injection and PDI side will take MBB. Second group takes the intervention in reverse order.

ELIGIBILITY:
Inclusion Criteria:

* CLBP of non-malignant origin fulfilling the following criteria:

  * Pain lasting for at least three months
  * Pain in both the left and right sides of the back
  * Pain below the L2 vertebral body
* Lumbar spine CT scan or MRI done in the last 2 years
* Average visual analogue scale (VAS) for pain ≥4/10 on each side for the 3 days
* Cognitive and physical ability to provide informed consent in English or French

Exclusion Criteria:

* Neurologic signs or symptoms suggesting nerve root involvement
* Strictly unilateral Low Back Pain (LBP)
* CT scan or MRI findings suggestive of pain etiology beyond degenerative spine disease

  * Vascular malformations
  * Tumor
  * Infection
  * Fractures
  * DISH (Diffuse idiopathic skeletal hyperostosis)
* Patients who have received injections of any type or acupuncture therapy to the low back in the last 3 months
* Prior spine surgery
* Local or systemic infection
* Bleeding disorder or the use of anticoagulation medications but for low-dose aspirin
* Known allergy to amid local anesthetics
* Active insurance claim (CSST, SAAQ)
* Uncontrolled psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-08; Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in Chronic Low Back Pain (CLBP) measured by VAS | Seven days

CONTACTS AND LOCATIONS:
Locations (1):
- Alan Edwards Pain Management Unit - Montreal General Hospital, Montreal, Quebec, Canada